CLINICAL TRIAL: NCT06361407
Title: Sensory and Cognitive Predictions, and Their Disruptions in Schizophrenia
Acronym: SensoSchiz
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Psychothérapique de Nancy (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-A02464-41
Record Dates: First submitted 2024-04-03; First posted 2024-04-11 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia; Sensory Processing Disorder
Keywords: sensory prediction; motion perception; prediction error
MeSH Terms: conditions — Schizophrenia | interventions — Neuropsychological Tests

STUDY DESIGN:
Intervention Model Description: Individuals with schizophrenia will be tested in parallel with neurotypicals
Masking Description: The group will be masked at the stage of data analysis. It cannot be masked at the prior stages
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- effect of trajectory perturbation (Experimental): All participants will run the task consisting in 2 squares moving towards each other. On each trial they will answer whether the squares touch or do not touch. All participants are tested with all experimental conditions. The rate of 'touch' responses will be compared when there is a trajectory perturbation without rebound vs. a trajectory with perturbation with rebound vs. a trajectory without perturbation and without rebound vs. a trajectory without perturbation and with rebound.
  Interventions: Behavioral: Illusion task

INTERVENTIONS:
Behavioral: Illusion task — The task is the illusion already described in the arm description. All participants will additionally benefit from a short neuropsychological evaluation exploring attention (CPT-AX) and semantic knowledge (fNART) and a clinical evaluation exploring the sense of self (EASE).
  Other Names: EASE evaluation; fNART; CPT-AX

SUMMARY:
Disturbances in the sense of self and time could play an important role in the development of psychotic symptoms. Previous work has shown that patients have difficulty preparing to process information on the scale of a second, but are abnormally disturbed by slightly asynchronous information on the millisecond scale. In both cases, the anomalies could explain the patients' unusual experience of time. The hypothesis in neurotypical patients is that small delays or asynchronies asynchronies are treated as irrelevant information and ignored and ignored, whereas in patients suffering from schizophrenia they would disrupt the flow of time. This hypothesis is tested with a new visual illusion.

DETAILED DESCRIPTION:
In the task, two squares move at constant speed in a straight line towards each other. When they collide and disappear neurotypical individuals perceive a gap between the two squares rather than contact. This unexpected effect cannot be explained by a 'cognitive' expectation, since what is consciously expected is collision and contact. It has been shown that it is sensory predictions which explain the illusion of space at the moment of contact. Indeed, a movement trajectory is accompanied by sensory predictions, which help to anticipate the position of the moving object, and of the contrast between the edges of the squares and the background. At the moment of collision, the contrast disappears and is processed as a prediction error. If subjects do not have time to correct the error, they see a gap, as if the figure-ground contrast was still there. Conversely, when a rebound effect is introduced into the task (the squares are moved in the opposite direction after the collision), the illusion diminishes, as if the rebound reinforces the (top-down) expectation of a collision.

Perturbations will be introduced during the trajectory in the illusion task with and without rebound to test this hypothesis (acceleration on a millisecond scale vs. uniform speed). Patients suffering from schizophrenia, whose prediction mechanisms are fragile, are expected to be abnormally sensitive to trajectory changes. The experimental manipulations will help to compare sensory prediction (illusion without rebound) and top-down (conscious) prediction (illusion with rebound).

The protocol will also help to specify which types of prediction (sensory or cognitive) underlie patients' sense patients' sense of self. In short, the protocol is designed to improve the pathophysiological understanding of sense-of-self disorders in schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Age between 18 and 60 inclusive;
* Subject having dated and signed the consent form prior to the start of any trial-related procedure (guardian or curator where applicable);
* Member of a social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* Psychoactive substance use disorders (as defined by the DSM-V) (Diagnostic and Statistical Manual-V);
* Use of benzodiazepines, hallucinogens (in the period preceding before inclusion, for a duration equivalent to 5 half-lives of the product) or cannabis (in the 2 months preceding inclusion);
* Neurological pathology or sequelae;
* Attention deficit hyperactivity disorder (ADHD);
* Borderline personality disorder;
* Disabling sensory disorders (visual acuity <0.8);
* Person deprived of liberty or under court protection;
* Pregnant, parturient or breast-feeding women;
* Subjects in a period of exclusion defined by another clinical study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Effect of a millisecond-level trajectory perturbation | Month 4
  Change in the rate of illusion in case of a trajectory perturbation (compared to the rate of illusion in the absence of perturbation)

SECONDARY OUTCOMES:
Baseline rate of illusion | month 4
  Frequency of the illusion perception when there is no trajectory perturbation and no rebound after the collision
Effect of a rebound (top-down, conscious influence) | month 4
  Change in the rate of illusion in case of a rebound (compared to the rate of illusion in the absence of rebound)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Giersch, MD PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France

IPD SHARING:
Plan to Share IPD: No